CLINICAL TRIAL: NCT03888963
Title: for Patients With Fibrocystic Disease of the Breast, Does Pulsed Radiofrequency on Thoracic Paravertebral Nerve Reduce Pain Severity
Brief Title: Pulsed Radiofrequency for Chronic Mastalgia of Fibrocystic Disease of the Breast
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Diab Fuad Hetta, Principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SECI-IRB-IORG0009563-726
Record Dates: First submitted 2019-03-22; First posted 2019-03-25 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF (Experimental)
  Interventions: Procedure: PRF
- SHAM (Sham Comparator)
  Interventions: Procedure: SHAM

INTERVENTIONS:
Procedure: PRF — patients will receive pulsed radiofrequency, 4 cycles (each cycle, 2 minutes) on the thoracic paravertebral nerves number 2,3, and 4 under fluroscopic guidance
  Arms: PRF
Procedure: SHAM — patients will be subjected to the same procedure like PRF group without giving PRF
  Arms: SHAM

SUMMARY:
The investigators will evaluate the analgesic efficacy of pulsed radiofrequency on the thoracic paravertebral nerves for patients with chronic mastalgia of fibrocystic disease of the breast

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic mastalgia due to fibrocystic disease of the breast
* the pain duration maintained for more than 1 year
* the pain intensity is more than 5 on VAS pain score

Exclusion Criteria:

* coagulopathy
* infection at the site of the procedure

Ages: 16 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-03-28 (Actual); Primary Completion 2019-08-20 (Estimated); Study Completion 2019-09-20 (Estimated)

PRIMARY OUTCOMES:
the changes in pain intensity measured by VAS pain score | patients will be evaluated at 3 months postoperatively
  VAS pain score, is a scale for pain measurements scored from 0 to 10 in which 0 = no pain and 10 = the worst imaginable pain

CONTACTS AND LOCATIONS:
Locations (1):
- Diab, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided